CLINICAL TRIAL: NCT04855279
Title: Effectiveness of Remineralization Agents on the Prevention of Dental Bleaching Induced Sensitivity
Brief Title: Prevention of Bleaching Induced Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Benin Dikmen, Assist. Prof. Dr., Medipol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KN453
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Tooth Bleaching; Tooth Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Glycerol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator)
  Interventions: Other: glycerine
- Topical neutral sodium fluoride (Active Comparator)
  Interventions: Other: neutral sodium fluoride
- ACP-CCP gel (Active Comparator)
  Interventions: Other: ACP-CCP gel
- nano-hydroxyapatite solution (Active Comparator)
  Interventions: Other: nano-hydroxyapatite solution

INTERVENTIONS:
Other: neutral sodium fluoride — Topically applied
  Arms: Topical neutral sodium fluoride
Other: ACP-CCP gel — Topically applied
  Arms: ACP-CCP gel
Other: nano-hydroxyapatite solution — Topically applied
  Arms: nano-hydroxyapatite solution
Other: glycerine — Topically applied
  Arms: Control

SUMMARY:
This study aims to evaluate the use of different desensitizing agents before in-office bleaching. A total of 64 volunteers were randomly divided into four groups. Before undergoing in-office bleaching with 38% hydrogen peroxide gel (three applications of 15 minutes each, one session), clinicians applied a placebo gel (control group), casein phosphopeptide-amorphous calcium phosphate (CPP-ACP), neutral sodium fluoride gel (NSF), or nano-hydroxyapatite solution (n-HAP) on all buccal surfaces of teeth. The gel was left undisturbed for 4 minutes. Patients recorded their tooth sensitivities on the VAS scale. Kruskal-Wallis test followed by Mann-Whitney U test were used to compare changes in tooth color and intensity of tooth sensitivity between groups.

DETAILED DESCRIPTION:
Color evaluation was performed with Vita Shade Guide Classical (Vitapan Classical, Vita, Bad Sakingen, Germany). The shades were evaluated with shade guide units (SGUs). Vita Classical Shade Guide consisted of 16 shades, and the shades were aligned light-to-dark from B1-C4.21, 22 The shades were taken before and after 24 hours and 7 days of treatment.Next, the hypersensitivity was recorded by asking each subject to establish his or her perception of sensitivity before treatment using a visual analog scale (VAS). A stimulus of an evaporative blowing triple syringe (25 psi at ambient conditions) was applied for 3 seconds on the upper central incisors from a distance of 1 cm. After 24 hours and 7 days of bleaching treatment, stimuli testing was performed again.The subjects were divided into four groups. Group 1. Subjects were treated with a placebo gel. The agent was applied for 4 min. to all the teeth to be bleached. Group 2. Subjects were treated with ACP-CCP gel (Tooth Mousse, GC Corp., Tokyo, Japan) for 4 min. to all the teeth to be bleached. Group 3. Subjects were treated with nano-hydroxyapatite solution for 4 min. to all the teeth to be bleached. Group 4. Subjects were treated with neutral sodium fluoride (NSF) gel for 4 min. to all the teeth to be bleached. After treatment, the agent was removed by washing with water in all groups. Each subject underwent one session of bleaching on the anterior teeth from canine-to-canine. Bleaching systems were applied according to the manufacturer's instructions by one of the authors. Subjects were treated with hydrogen peroxide at 38% activated by a light source composed of 12 LEDs with blue light generators. The calculated hypersensitivity values and color change values were tested with Shapiro-Wilk and Levene tests for normal data distribution and homogeneity of variances. Kruskal-Wallis test followed by Mann-Whitney U test was performed to compare groups.

ELIGIBILITY:
INCLUSION CRITERIA:

Must have all their upper and lower anterior teeth

Must have good oral hygiene

EXCLUSION CRITERIA:

Pregnancy or breastfeeding

Systemic disease

Taking NSAIDs or other drug treatment.

Periodontal disease

Enamel hypoplasia

Teeth stained by tetracycline or fluorosis

Dental malposition or orthodontic treatment with fixed appliances

Canine teeth lighter than A1

Restoration on anterior teeth

Cervical lesions

Symptoms of dental pain

Previous tooth whitening experience.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Effect of reducing hypersensitivity after bleaching | 1 week
  VAS scale (Visual Analog Scale) was measured before and after bleaching

CONTACTS AND LOCATIONS:
Overall Officials: Benin Dikmen, Dr., Principal Investigator — Medipol University
Locations (1):
- Medipol Mega University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reis A, Dalanhol AP, Cunha TS, Kossatz S, Loguercio AD. Assessment of tooth sensitivity using a desensitizer before light-activated bleaching. Oper Dent. 2011 Jan-Feb;36(1):12-7. doi: 10.2341/10-148-CR. Epub 2011 Mar 24. PMID 21488723